CLINICAL TRIAL: NCT06027450
Title: Bon USage Des ImmunoGlobulines Humaines Normales (IgHN) : Faisabilité de l'intégration Des critères de la hiérarchisation Lors Des Dispensations d'IgHN - BUS-IG
Brief Title: Good Use of Normal Human ImmunoGlobulins (NHIg): Feasibility of Integrating the Criteria of Hierarchy During of NHIg Dispensations
Acronym: BUS-IG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230354
Record Dates: First submitted 2023-08-21; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Immunoglobulins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with NHIg: Patients treated for one of the following indications :
  * Thrombopenic Idiopathic Purpura (TIP)
  * Chronic Demyelinating Inflammatory Polyradiculoneuritis (CDIP)
  * Secondary immune deficiency (SID)
  Interventions: Other: NHIg prescription

INTERVENTIONS:
Other: NHIg prescription — Analysis of NHIg prescription

SUMMARY:
Supply of Normal Human Immunoglobulins (NHIg) has been in steady tension for almost 15 years in the world. The scarcity of raw material, manufacturing time by industries, and increase consumptions are some of the causes. These phenomena has been accentuated for two years in the context of pandemic.

Faced these difficulties, the french National Medication Security Agency (ANSM) , in collaboration with health professionals and patients associations concerned, established a hierarchy of indications of NHIg to prioritize NHIg for patients without therapeutic alternative (2013 and 2019). Its use is sometimes complex, particularly in the indications where the use of NHIg must combine clinico-biological criteria and/or previous treatment lines.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with NHIg for one of the following 3 indications between 01/10/2021 and 31/12/2021: TIP, CDIP and SID.
* Patients 18 years of age and older

Exclusion Criteria:

* Patient Objection
* Patients treated with NHIg- for another indication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with NHIg for one of the following 3 indications between 01/10/2021 and 31/12/2021: TIP, CDIP and SID
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with clinical and biological information in the medical record | At inclusion
  * For TIP: Khellaf score present dating from less than a week
  * For CDIP: mention of at least one plasmapheresis since diagnosis and before NHIg prescription
  * For SID: mention of recent repeated infections (at least 2 infections that lead to hospitalization in the year before starting treatment) and rate of IgG dating from less than 3 months.

SECONDARY OUTCOMES:
Adequacy rate between NHIg indications noted in patients files and ANSM prioritization criteria | At inclusion
  * For TIP: Ig prescription if Khellaf score >8 dating from less than a week.
  * For CDIP: Ig prescription if plasmapheresis was executed in first intention
  * For SID: prescription of Ig if recent repeated infections (at least 2 infections that lead to hospitalization in the year before starting treatment) and rate of IgG dating from less than 3 months.
Number of patients prescribed treatment out of hierarchy | At inclusion
  Description of the criteria out of hierarchy, justifying the prescription of NHIg in these 3 authorized indications

IPD SHARING:
Plan to Share IPD: Undecided